CLINICAL TRIAL: NCT03015701
Title: Double Blind Randomized Trial of the Anti-Progestational Agent Mifepristone In The Treatment of Unresectable Meningioma
Brief Title: S9005 Mifepristone in Meningioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SWOG-9005; U10CA032102 (NIH)
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Meningioma
Keywords: Unresectable
MeSH Terms: conditions — Meningioma | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Mifepristone 200 mg orally daily for two years
  Interventions: Drug: Mifepristone
- Arm 2 (Placebo Comparator): Placebo orally daily for two years
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mifepristone — a 19 norsteroid with anti-progesterone and anti glucocorticoid activity which competitively inhibits binding of the hormone to its receptor
  Other Names: RU-486
  Arms: Arm 1
Other: Placebo — placebo matching mifepristone
  Arms: Arm 2

SUMMARY:
To compare daily oral mifepristone vs placebo with respect to time to treatment failure in patients with unresectable meningioma.

DETAILED DESCRIPTION:
To compare daily oral mifepristone vs placebo with respect to time to treatment failure in patients with unresectable meningioma and to address issues of safety in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically documented primary, recurrent or residual meningioma which is unresectable.
2. Patients must have active meningioma, which is defined to be one of the following:

   1. Progressive disease within the past 2 years.
   2. Recurrent Disease, as defined by the reappearance of a previously completely resected meningioma, within the past two years.
   3. New disease, defined as a diagnosis of meningioma within the previous two years
3. Patients must have measurable or evaluable disease which is documented on CT or MRI scan.
4. Patients should have already received radiotherapy unless radiotherapy is inappropriate due to tumor location(s) or unless radiotherapy, after discussion with the patient's physician, has been refused. If patients have received prior radiotherapy, this treatment must have been completed more than one year prior to study entry with documented progressive disease since completion of radiotherapy.
5. Patients must be 18 years or older, and must have a performance status 0-2 by Southwest Oncology Group criteria.
6. Patients must not have received prior cytotoxic chemotherapy for meningioma.
7. Patients must have serum creatinine, SGOT, and bilirubin ≤ 2 x IULN.
8. Patients requiring simultaneous administration of corticosteroids for cerebral edema must have been receiving a stable dose of corticosteroids for at least 4 weeks prior to study entry.
9. Patients receiving anti-epileptic medications are eligible. However barbiturates should be avoided if possible.
10. Patients with meningiomatosis (diffuse meningeal infiltration resulting in only nonevaluable meningeal thickening) are not eligible. However, patients with multiple measurable or evaluable meningioma tumor masses are eligible.
11. Patients with malignant meningioma are not eligible. Malignant meningioma is defined as meningioma that demonstrates hypercellularity, loss of architecture, nuclear pleomorphism, numerous mitoses, focal necrosis, and brain invasion.
12. Patients who have had additive or ablative modulation of sex hormone or glucocorticoid pathways within the preceding 3 months (not including stable corticosteroid therapy for cerebral edema) are not eligible. Such modulations include but are not limited to birth control pills, bilateral oophorectomy or orchiectomy, progestational inserts, oral or vaginal exogenous estrogens, androgens or antiandrogens, progestational agonists, tamoxifen, aminoglutethimide, o,p-DDD, ACTH, glucocorticoids not for cerebral edema, and leuprolides (or other LH-RH inhibitors). Patients must not have received prior mifepristone therapy for meningioma.
13. Patients must not have serious intercurrent medical illness; that is, any illness that in the opinion of the investigator would prevent following the study regimen.
14. Patients with clinical adrenal insufficiency requiring exogenous corticosteroid replacement are not eligible.
15. Patients with a known allergy to mifepristone are not eligible.
16. Patients with base of brain, cavernous sinus or optic nerve meningiomas or with visual symptoms must have a formal visual field examination.
17. Pregnant or lactating women may not participate. Pre-menopausal women and men of reproductive potential may not participate unless they have agreed to use an effective local contraceptive method (such as a condom, diaphragm, or IUD) or abstinence during and for 3 months after study therapy.
18. Patients with other prior or concurrent malignancy within the preceding 5 years, except surgically treated squamous or basal cell skin cancer or cervical cancer in situ, are not eligible.

    -

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 1992-08; Primary Completion 2001-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Time to Treatment Failure | 6 years
  From date of registration to first date of documentation of one of the following:
  1. Progression (clear worsening of evaluable disease must be confirmed by 2 investigators).
  2. Significant deterioration of at least one neurologic symptom
  3. Discontinuation of treatment for any reason.
  4. Death from any cause.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | two years after beginning treatment
  Patients will be followed for adverse events as defined by the SWOG toxicity criteria

CONTACTS AND LOCATIONS:
Overall Officials: Charles Blanke, MD, Study Director — Oregon Health and Sciences University

IPD SHARING:
Plan to Share IPD: Yes
https://swog.org/Visitors/Download/Policies/Policy43.pdf

REFERENCES:
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/